CLINICAL TRIAL: NCT02035007
Title: Transpulmonary Thermodilution Measurements in Patients With Heart Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version 2, 17.04.09 / EK1649
Record Dates: First submitted 2009-10-02; First posted 2014-01-14 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LV-EF > 50% (Experimental): PiCCO catheter analysis of patients with coronary heart disease without impaired left ventricular function [LV-EF > 50%]
  Interventions: Device: PiCCO Catheter (Pulsiocath 5F)

INTERVENTIONS:
Device: PiCCO Catheter (Pulsiocath 5F) — Measuring of PiCCO derived values
  Other Names: Pulsiocath 5F, Pulsion Medical Systems, Munich, Germany

SUMMARY:
The purpose of this study is to examine the validation of the PiCCO (Pulse Contour Cardiac Output)-derived transpulmonary thermodilution technology in patients with heart diseases.

DETAILED DESCRIPTION:
* How do PiCCO and PAC (pulmonary artery catheter) derived hemodynamic variables change in different cardiac pathologies?
* How do PiCCO hemodynamic variables compare to transthoracic echocardiographic parameters in different cardiac pathologies?
* How does GEDV (global enddiastolic volume) correlate with left ventricles end-diastolic volume (LVEDV) assessed by LV (left ventricle) ventriculography and echocardiography?
* How do PiCCO cardiac function variables (GEF [global ejection fraction]; CFI [cardiac function index]) correlate with LV dP/dt max, LVEF (left ventricular ejection fraction) assessed by LV ventriculography and echocardiography, LVFAC (left ventricular fractional area of change), LV stroke work index (LVSWI) and cardiac power (CP)?
* How does GEDV compare to LVEDV and left ventricular end-diastolic pressure (LVEDP) as assessed by the pulmonary artery occlusion pressure (PAOP)?
* How does right ventricular function influence GEDV, GEF and CFI?

ELIGIBILITY:
Inclusion criteria:

* Coronary heart disease without impaired left ventricular function [LV-EF > 50%] (n=10, control group)
* Coronary heart disease with impaired left ventricular function [LV-EF < 50%] (n=10)
* Dilated cardiomyopathy (n=10),
* Aortic valve stenosis (n=10),
* Mitral valve regurgitation (n=10),
* Diastolic left ventricular dysfunction (n=10) and
* Right heart failure (n=10)

Exclusion criteria:

* Patients with catecholamine dependent cardiogenic shock, severe respiratory distress because of pulmonary oedema, intubated patients, patients with atrial fibrillation, atrioventricular conduction abnormalities, and slow ventricular tachycardia will not be included.
* Moreover patients not being able to give informed consent are excluded. Even more, pregnant women are excluded from the study due to the radiation exposure in line with heart catheterization. A pregnancy test will be performed prior to participating with this study.
* The age does not represent an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cardiac Output, Preload values (GEDV) | Day 1 only
  Outcome measure is obtained during PiCCO measurement and left/right heart catherization, respectively ("point-of-care" measurement). There is no follow-up examination thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, Prof MD, Principal Investigator — University Hospital Zurich, Medical Intensive Care Unit
Locations (1):
- Medical Intensive Care Unit, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland